CLINICAL TRIAL: NCT06069908
Title: The Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Edema, Grip Strength, Dexterity and Quality of Life in Upper Extremity Lymphedema
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Upper Extremity Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seda Saka (Other)
Responsible Party: Sponsor-Investigator, Seda Saka, Associate Professor Doctor, Halic University
Organization: Halic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OzgeO
Record Dates: First submitted 2023-09-08; First posted 2023-10-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Quality of Life; Lymphedema; Hand Grasp; Grip; Strength; Edema
Keywords: Lymphedema; Hand Grip; Grip Strength; Quality of Life
MeSH Terms: conditions — Lymphedema; Edema | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Demographic data related to the patient will be questioned with the Demographic Data and Anamnesis form prepared by the researchers. Circumference measurement was determined as the primary outcome measure, and gross grip strength, dexterity and quality of life were determined as the secondary outcome measures. To this end; Patients' upper extremity circumference was measured with a tape measure, gross grip strength was measured with Jamar Dynanometer, manual dexterity was measured with 9-Hole Peg Test, upper extremity problems were measured with Arm, Shoulder and Hand Problems Quick Questionnaire (Quick DASH), items related to people's quality of life and specific arm symptoms were measured. Lymphedema Functionality will be evaluated with the Disability and Health Survey (LFÖSA) and quality of life will be evaluated with the Quality of Life Questionnaire in Upper Extremity Lymphedema Patients (ULL-27).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomly divided into three groups. Subjects will be instructed to draw an envelope from a secret box. Each envelope will contain a yellow, red and blue card and they will be assigned to one of the 3 groups of the study accordingly. Only the Complex Decongestive Treatment (manual lymph drainage, skin care, special exercises, compression) approach will be applied to the first group, Complex Decongestive Treatment and sham transcutaneous vagus nerve stimulation to the second group, and transcutaneous vagus nerve stimulation in addition to Complex Decongestive Treatment to the third group. The third party who has access to the box containing the envelopes will not be involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complex Decongestive Treatment (Placebo Comparator): Complex Decongestive Treatment (manual lymph drainage, skin care, special exercises, compression) approach. It will be applied 5 days a week for 3 weeks.
  Interventions: Other: Complex Decongestive Treatment; Other: Exercise
- Sham transcutaneous vagus nerve stimulation (Sham Comparator): In sham transcutaneous vagus nerve stimulation application, the device electrode will be placed in the superior scapha region of the outer ear, where the vagus nerve has no innervation, and no current will be given.Complex Decongestive Therapy and sham transcutaneous vagus nerve stimulation.It will be applied 5 days a week for 3 weeks.
  Interventions: Other: Complex Decongestive Treatment; Other: Sham transcutaneous vagus nerve stimulation; Other: Exercise
- Transcutaneous vagus nerve stimulation (Active Comparator): Transcutaneous vagus nerve stimulation will be applied in addition to Complex Decongestive Therapy.It will be applied 5 days a week for 3 weeks.
  Interventions: Other: Complex Decongestive Treatment; Other: Transcutaneous Auricular Vagus Nerve Stimulation; Other: Exercise

INTERVENTIONS:
Other: Complex Decongestive Treatment — Complex Decongestive Treatment (manual lymph drainage, skin care, special exercises, compression) approach. It will be applied 5 days a week for 3 weeks
Other: Sham transcutaneous vagus nerve stimulation — In sham transcutaneous vagus nerve stimulation application, the device electrode will be placed in the superior scapha region of the outer ear, where the vagus nerve has no innervation, and no current will be given.Complex Decongestive Therapy and sham transcutaneous vagus nerve stimulation.It will be applied 5 days a week for 3 weeks.
  Arms: Sham transcutaneous vagus nerve stimulation
Other: Transcutaneous Auricular Vagus Nerve Stimulation — Transcutaneous vagus nerve stimulation will be applied in addition to Complex Decongestive Therapy.It will be applied 5 days a week for 3 weeks.
  Arms: Transcutaneous vagus nerve stimulation
Other: Exercise — Patients will undergo lymphedema-specific exercises 5 days a week for 3 weeks.

SUMMARY:
Lymphedema is an inflammatory disease characterized by abnormal accumulation of excess water, plasma proteins, and extravascular blood and parenchymal cells in the affected upper and lower arms, chest and/or trunk due to inadequate lymphatic transport capacity, and is associated with high-severity, recurrent soft tissue infections that can lead to sepsis and even death. Although there is no definitive treatment for lymphedema, a Complex Decongestive Treatment approach that includes manual lymph drainage, skin care, special exercises, compression and personal care has been described to slow down the progression of the disease and prevent secondary complications. In addition, parasympathetic nerve activation has been described, similar to vagus nerve activation with manual lymphatic drainage. system activation can be increased. The aim of our study was to investigate the effect of transcutaneous auricular vagus nerve stimulation on quality of life, grip strength and manual dexterity in patients with unilateral upper extremity lymphedema. It was planned as a randomized controlled experimental study. The universe of the study will consist of lymphedema patients hospitalized in Gaziosmanpaşa Physical Therapy Rehabilitation Education and Research Hospital, and the sample will consist of 27 volunteer patients who meet the inclusion and exclusion criteria. The study was planned as a single-center (Gaziosmanpaşa Education and Research Hospital). Participants will be randomly divided into three groups. The groups will be determined by simple randomization method. Only Complex Decongestive Treatment (manual lymph drainage, skin care, special exercises, compression) approach will be applied to the first group, Complex Decongestive Treatment and sham transcutaneous vagus nerve stimulation will be applied to the second group, and transcutaneous vagus nerve stimulation will be applied in addition to Complex Decongestive Treatment to the third group. Data collected from the patients will be entered into SPSS 21.0 package program to create a data set and statistical analyses will be performed.

DETAILED DESCRIPTION:
Demographic data related to the patient will be questioned with the Demographic Data and Anamnesis form prepared by the researchers. Circumference measurement was determined as the primary outcome measure, and gross grip strength, dexterity and quality of life were determined as the secondary outcome measures. To this end; Patients' upper extremity circumference was measured with a tape measure, their gross grip strength was measured with the Jamar Dynanometer, manual skills were measured with the 9-Hole Peg Test, upper extremity problems were measured with the Arm, Shoulder and Hand Problems Quick Questionnaire (Quick DASH), items related to people's quality of life and specific arm symptoms were measured. Lymphedema Functionality will be evaluated with the Disability and Health Questionnaire (LFOSA) and the quality of life will be evaluated with the Quality of Life Questionnaire in Upper Extremity Lymphedema Patients (ULL-27).Upper Extremity Circumference Measurement will be evaluated for both upper extremities. Assuming the wrist pivot point, markings will be made every 4 cm up to the axilla. At the marked points, the circumference will be measured with a tape measure and the difference between the affected and healthy sides will be determined.The Jamar handheld dynamometer is the most reliable and most commonly used measuring tool for measuring static grip strength. Static and dynamic measurement dynamometers are used when evaluating grip strength. These devices are hydraulic, pneumatic, mechanical and resistive devices. Measurements are generally based on the principle of compressing two bars parallel to each other. Patients are positioned and evaluated according to the holding and grip strength of the dynamometer to be used. The needle of the Jamar Hand Dynamometer shows measurements up to a maximum of 90 kg. The person will be measured in a chair without arm support, with the arm in adduction and neutral rotation, the elbow in 90 degrees of flexion, and the forearm in a neutral position. Each measurement will be repeated three times, the average will be calculated and data will be created and recorded.The Nine-Hole Peg Test, which provides information about the functional status of the hand, consists of a board with nine holes and nine nails. While the test is applied to both hands, the application begins with the dominant hand. Before proceeding with the application part, the test procedure is read to the individuals who will perform the test. In the application part, individuals are asked to place the nails into the holes as soon as possible and to remove them without wasting time and place the nails in the empty chamber on the side. Meanwhile, the application time is measured using a stopwatch and recorded in seconds.The DASH scale is a criterion developed for the evaluation of disability related to the entire upper extremity and is used to monitor the level of disability and benefit from treatment. With the DASH scale, the difficulty encountered in performing 30 different activities related to the upper extremity in daily life is evaluated. The Quick-DASH survey used in this study is a survey created by selecting and organizing the 11 most used of these activities. Each question is evaluated at 5 levels and 1 point is given if the patient can do the activity without difficulty, and 5 points are given if the patient cannot do it at all. The results are calculated with the test's own formula. It is a questionnaire with proven validity and reliability in Turkish that measures physical functions and symptoms in patients with upper extremity problems.Lymphedema Functionality, Disability, and Health Questionnaire Devooogdt et al. It was developed by Kostanoğlu et al. in 2011, and its Turkish validity and reliability study was conducted by Kostanoğlu et al. in 2016. The survey consists of 29 questions. Each question is answered using a visual analog scale ranging from 0 - 100 mm. The questionnaire has five subdomains: physical function, mental function, home activities, mobility activities and social activities. The survey takes approximately 5 minutes to complete. The Lymphedema Functionality, Disability and Health Questionnaire will be administered to patients twice, before and after treatment.The reliability and validity of the ULL-27 questionnaire in upper extremity lymphedema due to breast cancer was conducted by Ayşe Kayalı in 2017. ULL-27 is a quality of life questionnaire consisting of 27 questions that considers upper extremity lymphedema as three components (physical, psychological and social components). The first 15 questions evaluate the physical component, questions between 16-22 evaluate the psychological component, and questions between 23-27 evaluate the social component. It is a 5-point Likert type scale (1 = strongly disagree, 5 = strongly agree). The lowest score is 27 and the highest score is 135. A high score from the scale indicates that lymphedema negatively affects the quality of life. The physical score consists of a total of fifteen questions and the person's score is between at least 15 and 75. The psychological score consists of seven questions with a minimum of 7 and a maximum of 35 points. There are five questions for the social score, with a minimum score of 5 and a maximum score of 25. For a total score of 27 questions, 1 of all questions will receive at least 27 points, and the person who chooses 5 of all questions will receive a maximum of 135 points.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Diagnosed with secondary lymphedema disease by the physician
* Minimum of three months after surgery
* Stage 2 and 3 patients
* Native speaker Turkish
* Individuals who agreed to participate in the study

Exclusion Criteria:

* Individuals with any neurological or orthopedic problems in the upper extremity
* Individuals undergoing upper extremity surgery
* Presence of cardiac edema
* Presence of arterial disease
* Presence of acute venous disease
* Those with sensory impairment
* Those with cardiac rhythm disorders
* Individuals with cooperation problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Extremity circumference measurement as the primary outcome measure | It will be evaluated before starting and at the end of treatment. It will take 3 weeks.
  Upper Extremity Circumference Measurement will be evaluated for both upper extremities. Assuming the wrist pivot point, markings will be made every 4 cm up to the axilla. The difference between the affected and healthy sides will be determined by measuring the circumference with a tape measure at the marked points.

SECONDARY OUTCOMES:
Gross grip strength | It will be evaluated before starting and at the end of treatment. It will take 3 weeks.
  Jamar hand dynamometer is the reliable and most commonly used measurement tool that measures static grip strength. Static and dynamic measurement dynamometers are used when evaluating grip strength. These devices are hydraulic, pneumatic, mechanical and resistive devices. Measurements are generally It is based on the principle of compressing two bars parallel to each other. Patients are positioned and evaluated according to the holding and grip strength of the dynamometer to be used. The needle of the Jamar Hand Dynamometer shows measurements up to a maximum of 90 kg.
  The person will be measured in a chair without arm support, with the arm in adduction and neutral rotation, the elbow in 90 flexion, and the forearm in neutral position. Each measurement will be repeated three times, the average will be calculated and data will be created and recorded.
Manual Dexterity | It will be evaluated before starting and at the end of treatment. It will take 3 weeks.
  The Nine-Hole Peg Test, which provides information about the functional status of the hand, consists of a board with nine holes and nine nails. While the test is applied to both hands, the application begins with the dominant hand. Before proceeding with the application part, the test procedure is read to the individuals who will perform the test. In the application part, individuals are asked to place the nails into the holes as soon as possible and to remove them without wasting time and place the nails in the empty chamber located on the side. Meanwhile, the application time is measured using a stopwatch and recorded in seconds.
Life Quality | It will be evaluated before starting and at the end of treatment. It will take 3 weeks.
  The Lymphedema Functioning, Disability and Health Questionnaire consists of 29 questions. Each question is answered using a visual analog scale ranging from 0 - 100 mm. The questionnaire has five subdomains: physical function, mental function, home activities, mobility activities and social activities. The survey takes approximately 5 minutes to complete. The Lymphedema Functioning, Disability and Health Survey will be administered to patients twice, before and after treatment. It is a quality of life survey consisting of 27 questions. It is a 5-point Likert type scale (1=strongly disagree, 5=strongly agree). The lowest score is 27 and the highest score is 135. A high score from the scale indicates that lymphedema negatively affects the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gümüşsu, MD, Study Director — Gaziosmanpaşa Eğitim ve Araştırma Hastanesi
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpaşa Training and Research Hospital, Istanbul, Gaziosmanpaşa
  - Halic University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capilupi MJ, Kerath SM, Becker LB. Vagus Nerve Stimulation and the Cardiovascular System. Cold Spring Harb Perspect Med. 2020 Feb 3;10(2):a034173. doi: 10.1101/cshperspect.a034173. PMID 31109966
- [Background] Cerritelli F, Frasch MG, Antonelli MC, Viglione C, Vecchi S, Chiera M, Manzotti A. A Review on the Vagus Nerve and Autonomic Nervous System During Fetal Development: Searching for Critical Windows. Front Neurosci. 2021 Sep 20;15:721605. doi: 10.3389/fnins.2021.721605. eCollection 2021. PMID 34616274
- [Background] de Sire A, Losco L, Lippi L, Spadoni D, Kaciulyte J, Sert G, Ciamarra P, Marcasciano M, Cuomo R, Bolletta A, Invernizzi M, Cigna E. Surgical Treatment and Rehabilitation Strategies for Upper and Lower Extremity Lymphedema: A Comprehensive Review. Medicina (Kaunas). 2022 Jul 19;58(7):954. doi: 10.3390/medicina58070954. PMID 35888673
- [Background] Drouin JS, Pfalzer L, Shim JM, Kim SJ. Comparisons between Manual Lymph Drainage, Abdominal Massage, and Electrical Stimulation on Functional Constipation Outcomes: A Randomized, Controlled Trial. Int J Environ Res Public Health. 2020 Jun 1;17(11):3924. doi: 10.3390/ijerph17113924. PMID 32492920
- [Background] Farmer AD, Strzelczyk A, Finisguerra A, Gourine AV, Gharabaghi A, Hasan A, Burger AM, Jaramillo AM, Mertens A, Majid A, Verkuil B, Badran BW, Ventura-Bort C, Gaul C, Beste C, Warren CM, Quintana DS, Hammerer D, Freri E, Frangos E, Tobaldini E, Kaniusas E, Rosenow F, Capone F, Panetsos F, Ackland GL, Kaithwas G, O'Leary GH, Genheimer H, Jacobs HIL, Van Diest I, Schoenen J, Redgrave J, Fang J, Deuchars J, Szeles JC, Thayer JF, More K, Vonck K, Steenbergen L, Vianna LC, McTeague LM, Ludwig M, Veldhuizen MG, De Couck M, Casazza M, Keute M, Bikson M, Andreatta M, D'Agostini M, Weymar M, Betts M, Prigge M, Kaess M, Roden M, Thai M, Schuster NM, Montano N, Hansen N, Kroemer NB, Rong P, Fischer R, Howland RH, Sclocco R, Sellaro R, Garcia RG, Bauer S, Gancheva S, Stavrakis S, Kampusch S, Deuchars SA, Wehner S, Laborde S, Usichenko T, Polak T, Zaehle T, Borges U, Teckentrup V, Jandackova VK, Napadow V, Koenig J. International Consensus Based Review and Recommendations for Minimum Reporting Standards in Research on Transcutaneous Vagus Nerve Stimulation (Version 2020). Front Hum Neurosci. 2021 Mar 23;14:568051. doi: 10.3389/fnhum.2020.568051. eCollection 2020. PMID 33854421
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Garcia Nores GD, Ly CL, Savetsky IL, Kataru RP, Ghanta S, Hespe GE, Rockson SG, Mehrara BJ. Regulatory T Cells Mediate Local Immunosuppression in Lymphedema. J Invest Dermatol. 2018 Feb;138(2):325-335. doi: 10.1016/j.jid.2017.09.011. Epub 2017 Sep 20. PMID 28942366
- [Background] Hilz MJ. Transcutaneous vagus nerve stimulation - A brief introduction and overview. Auton Neurosci. 2022 Dec;243:103038. doi: 10.1016/j.autneu.2022.103038. Epub 2022 Sep 27. PMID 36201901
- [Result] Ahmed U, Chang YC, Zafeiropoulos S, Nassrallah Z, Miller L, Zanos S. Strategies for precision vagus neuromodulation. Bioelectron Med. 2022 May 30;8(1):9. doi: 10.1186/s42234-022-00091-1. PMID 35637543